CLINICAL TRIAL: NCT00980889
Title: RCT Steel (Wallstent®) vs Nitinol (Wallflex®) Bile Duct Stent for Palliation of Malignant Obstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, claes soderlund, Stockholm South General Hospital, Stockholm South General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Steel vs nitinol
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Biliary Tract Neoplasms; Pancreatic Neoplasms; Stent Occlusion
Keywords: bile duct obstruction; jaundice; metal stent
MeSH Terms: conditions — Biliary Tract Neoplasms; Pancreatic Neoplasms; Cholestasis; Jaundice

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- steel (Active Comparator): Insertion of Metalic Steel Stent, Wallstent® in malignant distal bile duct obstruction
  Interventions: Device: Steel
- Nitinol (Active Comparator): Insertion of Metalic nitinol Stent, Wallflex® in malignant distal bile duct obstruction
  Interventions: Device: Nitinol

INTERVENTIONS:
Device: Steel — ERCP procedure insertion of Metalic Steel Stent, Wallstent®
  Other Names: Wallstent®
  Arms: steel
Device: Nitinol — Insertion of Metalic nitinol Stent, Wallflex® in malignant distal bile duct obstruction
  Other Names: Wallflex
  Arms: Nitinol

SUMMARY:
Less than 20% of patients with malignant distal bile duct (BD) obstruction (often pancreatic cancer) are suitable for resection surgery.In the rest,palliation treatment comes into focus. Jaundice caused by BD obstruction gives pain, infection (cholangitis), often itching and increased weight loss, and the patient is stigmatized by the deep yellow colour of the skin.Therefore palliation with endoscopic stenting by ERCP-technique is important. Modern self-expanding metal stents (SEMS) are now widely used in this context. Comparison in a RCT between steel and nitinol SEMS has never been performed.

The steel stent (Wallstent®) is the "original",is widely used, and has more expanding power. Nitinol stents are softer and claimed to be easier to insert,and are more and more popular.A newly developed nitinol stent (Wallflex®)may have these advantages, but is some 120 Euros more expensive.

Regarding the most important outcome measure, time to stent failure (obstruction), no one knows if there is any difference.Our hypothesis is that there is no difference in this main outcome endpoint.

DETAILED DESCRIPTION:
Secondary outcome measures (compare above) are complications caused by the stent or stent insertion and technical ease to insert the stent. To discover a 12% difference between the 2 groups, regarding patency, 400 patients must be included in the trial, alfa 0.05, beta 0.8. Investigators know from previous trials (Single center trial South Hospital GIE 2006;63:986-995 and a newly finished similar swedish multicenter trial,prel data DDW- 09)that the 9 hospitals recruited will be able to include this no of patients in approximately 2.5 years.

Investigators will have a shortest follow-up period of 10 months, followup will be by phone with standard questions connected to stent failure, which is defined clinically AND by a new ERCP with intervention because of an obstructed stent.

ELIGIBILITY:
Inclusion Criteria:

* pt more than 20yrs.
* BD stenosis at least 2cm distal of the hepatic hilum, with typical malignant exposure radiologically.
* Clinically in accordance with tumour.s-bilirubin more than 50 micromol per litre.
* Radical surgery probably not possible(temporary-1month-plastic stenting for further investigation and then exchange to SEMS if estimated non-operable, after Rx is allowed).
* The patient must be fully informed by his doctor orally and in writing prior to the procedure, and give her/his informed consent. Ultrasound or CT examination must be performed prior to Rx.

Exclusion Criteria:

* Informed consent not obtained.
* Significant multiple intrahepatic stenosis by multiple tumour growth, not suitable for ERCP stenting.
* Radical Surgery will probably take place. Suspicion of non-malignant obstruction-further investigation must be performed.
* Not possible by anatomical reasons to reach the papilla, i.e because of prior operations.

prior BD stent inserted (metal stent or plastic stent >1month).

* Previously included in this trial. Prothrombin index more than 1.5. (normal <1.1).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
confirmed stent failure | 300 days follow up

SECONDARY OUTCOMES:
safety with respective stent in trial at insertion and afterwards(complic.) | 300 days
Survival | 300 days
  Survival difference between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Claes soderlund, assist prof, Principal Investigator — south hospital, stockholm sweden
Locations (11):
- Sweden (11):
  - Department of Surgery, Upper GI Div. South Hospital,, Stockholm, SLL
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Länssjukhuset Ryhov, Jönköping
  - Länssjukhuset i Kalmar, Kalmar
  - Blekingesjukhuset, Karlskrona
  - Centralsjukhuset i Kristianstad, Kristianstad
  - Universitetssjukhuset i Lund, Lund
  - Universitetssjukhuset i Malmö,, Malmo
  - dept surgery, South Hospital-Karolinska Institute, Stockholm
  - Claes.Soderlund, Stockholm
  - Vasteraslasarett, Västerås

REFERENCES:
- [Derived] Soderlund C, Linder S, Bergenzaun PE, Grape T, Hakansson HO, Kilander A, Lindell G, Ljungman M, Ohlin B, Nielsen J, Rudberg C, Stotzer PO, Svartholm E, Toth E, Frozanpor F. Nitinol versus steel partially covered self-expandable metal stent for malignant distal biliary obstruction: a randomized trial. Endoscopy. 2014 Nov;46(11):941-8. doi: 10.1055/s-0034-1377936. Epub 2014 Oct 16. PMID 25321620